CLINICAL TRIAL: NCT06373484
Title: Matching Assessment and Treatment for Children With Disruptive Behaviour and Their Parents
Acronym: MATCH-DB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018-2022
Record Dates: First submitted 2024-01-17; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Disruptive Behavior Disorder; Emotional Disorder; Behavioural Disorder; Attention Deficit Hyperactivity Disorder; Conduct Disorder; Oppositional Defiant Disorder
Keywords: Emotional and Behavioural Disorders; Disruptive Behaviour Disorder; Attention Deficit Hyperactivity Disorder; Conduct Disorder; Oppositional Defiant Disorder; Parenting Skills; Behavioural Parenting Training
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Mental Disorders; Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Component Child and Parent Cognitive Behavioral Therapy (Experimental): Parents and their children aged 6-12 with DBD who meet inclusion criteria.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Two 15-session multi-component cognitive-behavioral group treatments for children with disruptive behavior and their parents (i.e., one program for children aged 6-8 years and their parents and another for children aged 9-12 years and their parents. The programs have a child and parent group that are implemented concurrently).

SUMMARY:
This study will develop and test whether personalized profiles of children with Disruptive Behaviour Disorder (DBD) and their parents based on important psychological, emotional, and neuropsychological indicators predict their response to child cognitive behavioral treatment and Behavioral Parent Training.

DETAILED DESCRIPTION:
To accomplish these goals, the investigators will collect psychological, emotional, and neuropsychological measures before and following cognitive behavioural therapy (CBT) for both children and parents. The investigators will use statistical modeling to determine profiles of parents of children and children aged 6-12 years with DBD based on key domains of mental health, emotion regulation, cognition, and parent-child behaviour, and observe whether these profiles allow the study team to predict which sub-groups of parents and children are most and least likely to benefit from child CBT and Behavioural Parent Training (BPT).

ELIGIBILITY:
Inclusion Criteria:

* Child is borderline/clinically at risk on the Child Behaviour Checklist (CBCL) or Teacher Report Form (TRF) (T-score greater than or equal to 60 on Externalizing Problems composite scale or a T-score greater than or equal to 65 on the Oppositional Defiant Disorder and/or Conduct Disorder scales)
* Child has clinically severe impairment in the interpersonal relations (greater than 3), functioning in schoolwork (greater than 3), or total domains (greater than 15) on the Columbia Impairment scale.
* Parent is able and willing to participate in a group treatment

Exclusion Criteria:

* Child has an ongoing query or diagnosis of Pervasive Developmental Disorder or Autism or Asperger's Disorder
* Evidence of cognitive delays or an intellectual disability (based on the Kauffman Brief Intelligence Test-2 (KBIT-2), verbal and/or IQ composite standard score below 80 or collateral information)
* Child behaviour or emotional functioning that make group participation not possible
* Child preference for individual treatment.
* Parent behaviour or emotional functioning that make group participation not possible
* Parent preference for individual treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Changes in parenting skills between baseline, post-treatment, and follow-up (6 months - 1 year) | Baseline and post-treatment and follow-up (6 months - 1 year)
  Parenting skills are assessed using the Alabama Parenting Questionnaire (APQ). Parents indicate how often an item typically occurs in their home: 'never', 'almost never', 'sometimes', 'often', or 'always'.
Changes in parenting competencies between baseline, post-treatment, and follow-up (6 months - 1 year) | Baseline and post-treatment and follow-up (6 months - 1 year)
  Parenting competencies are assessed using the Parenting Sense of Competence (PSOC). Parents indicate how much they agree with statements: 'strongly disagree', 'disagree', 'slightly disagree', 'slightly agree', 'agree', or 'strongly agree'.
Changes in child emotional and behavioral problems between baseline, post-treatment, and follow-up (6 months - 1 year) | Baseline and post-treatment and follow-up (6 months - 1 year)
  Child emotional and behavioral problems are assessed using the Strengths and Difficulties Questionnaire (SDQ), Behavior and Feelings Scale (BFS), Child Behavior Checklist (CBCL), and the Modified Connors. The SDQ asks asks parents to indicate how true a statement is with regards to their child's emotions or behaviours in the last 6 months: 'not true', 'somewhat true', or 'certainly true'. The BFS asks parents to indicate how big of a problem a behaviour or feeling has been for a child in the last two weeks from '0 - not a problem' to '4 - a very big problem'. The CBCL asks parents to indicate how relevant the listed challenges are to their child from '0 - not true', '1 - somewhat or sometime true', and '2 - very or often true'. The Modified Connors asks parents to indicate how much a concerning behaviour describes their child from 'not at all', 'just a little', 'pretty much', or 'very much'.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan F. Andrade, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available following publication for up to one year.
Access Criteria: Information will be shared with qualified investigators at the discretion of the principal investigator.

REFERENCES:
- [Background] Andrade BF, Sorge GB, Na JJ, Wharton-Shukster E. Clinical Profiles of Children with Disruptive Behaviors Based on the Severity of Their Conduct Problems, Callous-Unemotional Traits and Emotional Difficulties. Child Psychiatry Hum Dev. 2015 Aug;46(4):567-76. doi: 10.1007/s10578-014-0497-8. PMID 25257946
- [Background] Aitken M, Waxman JA, MacDonald K, Andrade BF. Effect of Comorbid Psychopathology and Conduct Problem Severity on Response to a Multi-component Intervention for Childhood Disruptive Behavior. Child Psychiatry Hum Dev. 2018 Dec;49(6):853-864. doi: 10.1007/s10578-018-0800-1. PMID 29594940
- [Background] Ludmer JA, Sanches M, Propp L, Andrade BF. Comparing the Multicomponent Coping Power Program to Individualized Parent-Child Treatment for Improving the Parenting Efficacy and Satisfaction of Parents of Children with Conduct Problems. Child Psychiatry Hum Dev. 2018 Feb;49(1):100-108. doi: 10.1007/s10578-017-0732-1. PMID 28500434
- [Background] Leijten P, Gardner F, Landau S, Harris V, Mann J, Hutchings J, Beecham J, Bonin EM, Scott S. Research Review: Harnessing the power of individual participant data in a meta-analysis of the benefits and harms of the Incredible Years parenting program. J Child Psychol Psychiatry. 2018 Feb;59(2):99-109. doi: 10.1111/jcpp.12781. Epub 2017 Jul 11. PMID 28696032
- [Background] Lochman, J.E. and K.C. Wells, Effectiveness of the Coping Power Program and of Classroom Intervention With Aggressive Children: Outcomes at a 1-Year Follow-Up. Behavior Therapy, 2003. 34: p. 493-515.
- [Background] Andrade, B.F., et al., The clinic adapted coping power program compared to individualized treatment; A randomized and controlled efficacy trial. 2018. In Progress.
- [Background] Lochman, J.E. and K.C. Wells, Effectiveness of the Coping Power Program and of classroom intervention with aggressive children: Outcomes at 1-year follow-up. Behavior Therapy, 2003. 34(4): p. 493-515.
- [Background] Andrade, B.F., et al., The clinic-adapted coping power program and individualized child and family treatment: A randomized and controlled effectiveness trial. In preparation, 2015.
- [Background] Andrade, B.F., et al., Implementation and evaluation of an evidence-based treatment for disruptive behaviour within a children's mental health program. Canadian Journal of Program Evaluation, 2015. 2015, 30(2): p. 195-204.
- [Background] Kil H, Aitken M, Henry S, Hoxha O, Rodak T, Bennett K, Andrade BF. Transdiagnostic Associations Among Parental Causal Locus Attributions, Child Behavior and Psychosocial Treatment Outcomes: A Systematic Review. Clin Child Fam Psychol Rev. 2021 Jun;24(2):267-293. doi: 10.1007/s10567-020-00341-1. Epub 2021 Feb 18. PMID 33598852